CLINICAL TRIAL: NCT01325649
Title: Optimal Surgery With Total Mesorectal Excision and MRI Based Multimodal Therapy of Rectal Carcinoma
Brief Title: Optimal Surgery and MRI Based Radiochemotherapy in Rectal Carcinoma
Acronym: OCUM
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Theo Junginger, MD, Johannes Gutenberg University Mainz
Other Study IDs: Ocumstudy 19.08.2009
Record Dates: First submitted 2011-03-28; First posted 2011-03-30 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Rectal Cancer Stage II; Rectal Cancer Stage III
Keywords: rectal cancer; MRI; selective preoperative radiochemotherapy; involvement of circumferential resection margin; locoregional recurrence rate
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- advanced rectal cancer: Patients with carcinoma of the middle rectum with positive mrCRM (≤ 1 mm), with cT3 low rectal carcinoma, and with cT4 Tumors Arm 1 Long course radiochemotherapy before total mesorectal excision Arm 2 total mesorectal excision without radiochemotherapy
  Interventions: Procedure: total mesorectal excision / long course radiochemotherapy; Radiation: long course 5-FU bases radiochemotherapy

INTERVENTIONS:
Procedure: total mesorectal excision / long course radiochemotherapy — long course 5-FU based radiochemotherapy before total mesorectal excision
Radiation: long course 5-FU bases radiochemotherapy

SUMMARY:
The objective of the study is to provide proof that a MRI based preoperative radiochemotherapy in patients with locally advanced rectal carcinoma allows limiting RCT to high risk patients without increase of locoregional recurrence rate and decrease of overall survival provided there is a high quality of mesorectal excision.

DETAILED DESCRIPTION:
The criteria for application of RCT is the distance of the tumor from mesorectal fascia in preoperative MRI of the pelvis. In case of a T 4 tumor or a tumor with a distance of 1mm of less form mesorectal fascia long-course radiochemotherapy is applied followed by surgery, in all other cases primary surgery is done.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed invasive carcinoma of the rectum infiltrating beyond the submucosa (cT3, cT2N+, cM0)
* Elective surgery
* Fit for surgery
* Preoperative MRI of pelvis

Exclusion Criteria:

* uT1 Tumors
* provided for local excision
* previous or synchronous malignant tumors (except squamous and basal cell carcinoma of the skin and carcinoma in situ of the cervix)
* previous irradiation of the pelvis
* ulcerative colitis or Crohn's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with carcinoma of the middle rectum with positive mrCRM (≤ 1 mm), with cT3 low rectal carcinoma, and with cT4 tumors
Sampling Method: Non-Probability Sample
Enrollment: 1051 (Actual)
Dates: Start 2009-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Locoregional recurrence rate | Five year

SECONDARY OUTCOMES:
Rate of involvement of circumferential resection margin (pCRM positive of resected specimens | postoperative
  pCRM positive means a distance of the tumor from circumferential resection margin 1mm or less.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medicine Center Department of General and Abdomial Surgery, Mainz, Germany

REFERENCES:
- [Derived] Ruppert R, Junginger T, Kube R, Strassburg J, Lewin A, Baral J, Maurer CA, Sauer J, Lauscher J, Winde G, Thomasmeyer R, Stelzner S, Bambauer C, Scheunemann S, Faedrich A, Wollschlaeger D, Merkel S. Risk-Adapted Neoadjuvant Chemoradiotherapy in Rectal Cancer: Final Report of the OCUM Study. J Clin Oncol. 2023 Aug 20;41(24):4025-4034. doi: 10.1200/JCO.22.02166. Epub 2023 Jun 19. PMID 37335957
- [Derived] Ruppert R, Kube R, Strassburg J, Lewin A, Baral J, Maurer CA, Sauer J, Junginger T, Hermanek P, Merkel S; other members of the OCUM Group. Avoidance of Overtreatment of Rectal Cancer by Selective Chemoradiotherapy: Results of the Optimized Surgery and MRI-Based Multimodal Therapy Trial. J Am Coll Surg. 2020 Oct;231(4):413-425.e2. doi: 10.1016/j.jamcollsurg.2020.06.023. Epub 2020 Jul 19. PMID 32697965
- [Derived] Kreis ME, Ruppert R, Ptok H, Strassburg J, Brosi P, Lewin A, Schon MR, Sauer J, Junginger T, Merkel S, Hermanek P; OCUM study group. Use of Preoperative Magnetic Resonance Imaging to Select Patients with Rectal Cancer for Neoadjuvant Chemoradiation--Interim Analysis of the German OCUM Trial (NCT01325649). J Gastrointest Surg. 2016 Jan;20(1):25-32; discussion 32-3. doi: 10.1007/s11605-015-3011-0. Epub 2015 Nov 10. PMID 26556476
- [Derived] Kreis ME, Maurer CA, Ruppert R, Ptok H, Strassburg J, Junginger T, Merkel S, Hermanek P. [Lymph node dissection after primary surgery and neoadjuvant radiochemotherapy of rectal cancer. Interim analysis of a multicenter prospective observational study (OCUM)]. Chirurg. 2015 Dec;86(12):1132-7. doi: 10.1007/s00104-015-0062-4. German. PMID 26223668